CLINICAL TRIAL: NCT02558751
Title: Immune Response to Pneumococcal Vaccination in Aging HIV Positive Individuals
Brief Title: Pneumonia Vaccine in Aging HIV Positive Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AG045973 (NIH); R01AG045973 (NIH)
Record Dates: First submitted 2015-09-16; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Pneumococcal Infection
Keywords: pneumococcal conjugate vaccine; aging HIV
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIV positive PPV23 (Active Comparator): HIV-positive individuals 50-65 years of age immunized with one dose of the 23-valent pneumococcal polysaccharide vaccine, PPV23
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- HIV positive PCV13/PPV23 (Active Comparator): HIV-positive individual 50-65 years of age, Intervention: one dose of 13-valent pneumococcal conjugate vaccine,PCV13, followed 8 weeks later with one dose of 23-valent pneumococcal polysaccharide vaccine, PPV23
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: 13-valent pneumococcal conjugate vaccine
- HIV negative PCV13/PPV23 (Active Comparator): HIV-negative individual 50-65 years of age, Intervention: one dose of 13-valent pneumococcal conjugate vaccine,PCV13, followed 8 weeks later with one dose of 23-valent pneumococcal polysaccharide vaccine, PPV23
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 23-valent pneumococcal polysaccharide vaccine — One standard adult dose of the 23-valent pneumococcal polysaccharide vaccine
  Other Names: PPV23 or Pneumovax
Biological: 13-valent pneumococcal conjugate vaccine — One dose of the 13-valent pneumococcal conjugate vaccine, PCV13, followed 8 weeks later by one dose of the 23-valent pneumococcal polysaccharide vaccine, PPV23.
  Other Names: PCV13 or Prevnar 13
  Arms: HIV negative PCV13/PPV23; HIV positive PCV13/PPV23

SUMMARY:
The investigators hypothesized that vaccination with either the 23-valent pneumococcal polysaccharide vaccine (PPV23) alone or the 13-valent pneumococcal conjugate vaccine (PCV 13) followed by PPV23 results in similar antibody levels/functional activity and induce a similar pneumococcal polysaccharide (PPS)-specific B cell response in HIV-positive individuals >50 years of age and HIV-negative persons>50 years of age. The investigators immunized the study group HIV+ persons>50 and controls (HIV negative >50 years) with PCV13 followed by PPV23 and HIV+>50 with PPV23 alone. The investigators examined immune responses to PPS23F and PPS14 on a quantitative and qualitative level using ELISA and opsonophagocytic assays (OPA).

To test the hypothesis that the levels of antigen specific B cells identified with PPS were comparable between the PPV23 and PCV13 vaccine recipients. Pre- and post-immunization peripheral blood samples were obtained. Extensive B cell phenotype analysis using fluorescent antibodies was used to characterize PPS-labeled B cells. Specific phenotypes were correlated with antibody levels and OPA and compared to historic populations immunized with PPV.

DETAILED DESCRIPTION:
All potential study candidates were asked to fill out a questionnaire concerning their medical history and medications. This survey determined eligibility. If eligible, as part of the experimental protocol the HIV positive participants agreed to be randomized to PPV23 alone versus PCV13 followed 8 weeks later by PPV23 immunization and 3 to 5 blood draws around the time of immunization. The HIV negative control population agreed to immunization with PCV13 followed 8 weeks later by PPV23, not standard of care for this population, and 5 blood draws around the time of immunization. The investigators compared the effect of single dose pneumococcal polysaccharide vaccination versus PCV13 followed by PPV23 vaccination in HIV positive adults. Prior to 2012, the standard of care of HIV positive adults included vaccination with PPV23. In 2012, these recommendations changed and it was recommended that all HIV positive adults be vaccinated with PCV13 followed at least 8 weeks later by PPV23. The benefit of this vaccination protocol over PPV23 alone in HIV positive adults >50 years of age however had not been studied. As part of this study, all HIV positive adults>50 years of age and a CD4 count>200 who were due for pneumococcal vaccination as standard of care, were asked to participate in the study. Those who agreed and were eligible to participate were randomly assigned to receive PCV13 followed at least 8 weeks later with PPV23 or received a single vaccination with PPV23. As standard of care, all individuals who were due for their pneumococcal vaccine and were not eligible for the study received PCV13 followed by PPV23.

The HIV positive volunteers (n=37) agreed to (experimental part of the protocol):

1. Be randomized to either vaccination with PCV13 followed by PPV23 OR PPV23 alone.
2. Donate blood specimens at 3-5 different times:

   PPV23 group:day 0, day of vaccination: 2 mL, at day 7, 40 mL and at day 28-42 a one time sample of 2 mL PCV13/PPV23 group: day 0, day of vaccination with PCV13: 2 mL, at day 7, 40 mL and at day 56, day of PPPV23, 2 mL, day 63 a 40 mL sample and finally at day 90 a one time sample of 2 mL.
3. Have blood samples subjected to antibody analysis (concentration and functional activity) and PPS-specific B cell phenotype and tumor necrosis factor receptors (TNFR) .

The HIV negative controls in the study (n=14) who agree to participate were vaccinated with the PCV13 followed by PPV23.This is NOT a vaccine regime recommended for healthy adults but is NOT contraindicated.

Thus as part of the experimental procedure for these individuals they will:

1. Receive the FDA approved PCV13 and PPV23
2. Blood samples were obtained at day 0, day of vaccination with PCV13: 2 mL, at day 7, 40 mL and at day 56, day of PPPV23, 2 mL, day 63 a 40 mL sample and finally at day 90 a one time sample of 2 mL.
3. Blood samples were analyzed for antibody concentration, functional activity and PPS-specific B cell phenotype and TNFR.

In summary,the investigators studied 3 populations, all were between 50-65 years of age:

Group 1: HIV positive CD4>200 vaccinated with PPV23 Group 2: HIV positive CD4> 200 vaccinated with PCV13 followed 8 weeks later by PPV23 Group 3: HIV negative vaccinated with PCV13/PPV23.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative:
* never immunized with PCV13
* HIV positive:
* need for pneumococcal vaccination per standard of care

Exclusion Criteria:

* steroid use
* other immunosuppressive agents;
* pregnancy
* incapable of completing consent form

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Antibody response measured by ELISA (ug/ml) | Change in ug/ml from day 0 to day 30
Opsonophagocytic antibody activity measured by opsonophagocytic assay (OPA titer) | Change in OPA titer from day 0 to day 30
Antibody response measured by ELISA (ug/ml) | Change in ug/ml from day 0 to day 90
Opsonophagocytic antibody activity measured by opsonophagocytic assay (OPA titer) | Change in OPA titer from day 0 to day 90

SECONDARY OUTCOMES:
B cell phenotype of PPS-specific B cells expressing CD27+IgM+: flowcytometry (%) | Change from day 0 to day 7 in %
Serum C-reactive protein (ng/ml) | day 0
Flow cytometry : percentage cells expressing BAFF-R on surface (%) | Change from day 0 to day 7
Flow cytometry : percentage cells expressing BAFF-R on surface (%) | Change from day 56 to day 63
B cell phenotype of PPS-specific B cells expressing CD27IgM: flowcytometry (%) | Change from day 56 to day 63 (%)
Serum IL-6 level (pg/ml) | Day 0
Serum sCD27 (U/ml) | Day 0
Serum sCD30 (U/ml) | Day 0
Serum BAFF concentration (pg/ml) | Day 0
Serum TACI concentration (pg/ml) | Day 0
Serum BCMA concentration (pg/ml) | Day 0
Flow cytometry : percentage cells expressing CD40 on surface (%) | Change from day 0 to day 7 (%)
Flow cytometry : percentage cells expressing CD40 on surface (%) | Change from day 56 to day 63 (%)
Flow cytometry : percentage cells expressing CD21 on surface (%) | Change from day 0 to day 7 (%)
Flow cytometry : percentage cells expressing CD21 on surface (%) | Change from day 56 to day 63 (%)
Flow cytometry : percentage cells expressing TACI on surface (%) | Change from day 0 to day 7 (%)
Flow cytometry : percentage cells expressing TACI on surface (%) | Change from day 56 to day 63 (%)

CONTACTS AND LOCATIONS:
Overall Officials: Maria AJ Westerink, M.D., Principal Investigator — University of Toledo
Locations (1):
- The University of Toledo-Health Science Campus, Toledo, Ohio, United States

REFERENCES:
- [Result] Ballet JJ, Sulcebe G, Couderc LJ, Danon F, Rabian C, Lathrop M, Clauvel JP, Seligmann M. Impaired anti-pneumococcal antibody response in patients with AIDS-related persistent generalized lymphadenopathy. Clin Exp Immunol. 1987 Jun;68(3):479-87. PMID 3652522
- [Result] Janoff EN, Douglas JM Jr, Gabriel M, Blaser MJ, Davidson AJ, Cohn DL, Judson FN. Class-specific antibody response to pneumococcal capsular polysaccharides in men infected with human immunodeficiency virus type 1. J Infect Dis. 1988 Nov;158(5):983-90. doi: 10.1093/infdis/158.5.983. PMID 3183430
- [Result] Klein RS, Selwyn PA, Maude D, Pollard C, Freeman K, Schiffman G. Response to pneumococcal vaccine among asymptomatic heterosexual partners of persons with AIDS and intravenous drug users infected with human immunodeficiency virus. J Infect Dis. 1989 Nov;160(5):826-31. doi: 10.1093/infdis/160.5.826. PMID 2572650
- [Result] Kroon FP, van Dissel JT, Ravensbergen E, Nibbering PH, van Furth R. Enhanced antibody response to pneumococcal polysaccharide vaccine after prior immunization with conjugate pneumococcal vaccine in HIV-infected adults. Vaccine. 2000 Nov 22;19(7-8):886-94. doi: 10.1016/s0264-410x(00)00232-2. PMID 11115712
- [Result] Rodriguez-Barradas MC, Musher DM, Lahart C, Lacke C, Groover J, Watson D, Baughn R, Cate T, Crofoot G. Antibody to capsular polysaccharides of Streptococcus pneumoniae after vaccination of human immunodeficiency virus-infected subjects with 23-valent pneumococcal vaccine. J Infect Dis. 1992 Mar;165(3):553-6. doi: 10.1093/infdis/165.3.553. PMID 1347058